CLINICAL TRIAL: NCT01681472
Title: A Single-Blind, Randomized Phase I/II Study of Pharmacokinetic and Pharmacodynamic Investigation of Modufolin® (60 or 200mg/m2) Compared to Levoleucovorin (60 or 200mg/m2) in Tumor, Adjacent Mucosa and Plasma for Patients With Colon Cancer
Brief Title: PK/PD Investigation of Modufolin (Arfolitixorin) in Plasma, Tumor and Adjacent Mucosa Adjacent Mucosa in Patients With Colon Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isofol Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISO-CC-002; 2012-000522-22 (EudraCT Number)
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Results first posted 2015-07-17 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Colonic Neoplasms
Keywords: Colon cancer; 5,10-methylenetetrahydrofolate; Rectal Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases; Therapeutic Uses; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases | interventions — 5,10-methylenetetrahydrofolic acid; Levoleucovorin; Leucovorin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Levoleucovorin 200 mg/m2 (Active Comparator): One i.v. bolus injection of study drug after the patient has been anaesthetized.
  Interventions: Drug: Levoleucovorin 200 mg/m2
- Levoleucovorin 60 mg/m2 (Active Comparator): One i.v. bolus injection of study drug after the patient has been anaesthetized.
  Interventions: Drug: Levoleucovorin 60 mg/m2
- 6R-MTHF 200 mg/m2 (Experimental): One i.v. bolus injection of study drug after the patient has been anaesthetized.
  Interventions: Drug: 6R-MTHF (arfolitixorin) 200 mg/m2
- 6R-MTHF 60 mg/m2 (Experimental): One i.v. bolus injection of study drug after the patient has been anaesthetized.
  Interventions: Drug: 6R-MTHF (arfolitixorin) 60 mg/m2

INTERVENTIONS:
Drug: 6R-MTHF (arfolitixorin) 200 mg/m2 — i.v. bolus injection
  Other Names: Modufolin®; ISO-901; [6R] 5,10-methylenetetrahydrofolate; arfolitixorin
  Arms: 6R-MTHF 200 mg/m2
Drug: Levoleucovorin 200 mg/m2 — i.v. bolus injection
  Other Names: Isovorin®
  Arms: Levoleucovorin 200 mg/m2
Drug: 6R-MTHF (arfolitixorin) 60 mg/m2 — i.v. bolus injection
  Other Names: Modufolin®; ISO-901; [6R] 5,10-methylenetetrahydrofolate; arfolitixorin
  Arms: 6R-MTHF 60 mg/m2
Drug: Levoleucovorin 60 mg/m2 — i.v. bolus injection
  Other Names: Isovorin®
  Arms: Levoleucovorin 60 mg/m2

SUMMARY:
The purpose of this study is to compare the concentration of four different metabolites in the tumor, in adjacent mucosa and in plasma in patients with colon cancer receiving two different doses of Modufolin (arfolitixorin) and Levoleucovorin (Isovorin®), respectively (60 and 200 mg/m2).

DETAILED DESCRIPTION:
The purpose of this study is to compare the concentration of [6R] 5,10-methylene-THF, 5-formyl-THF, 5-methyl-THF and THF in the tumor, in adjacent mucosa and in plasma in patients with colon cancer receiving two different does of Modufolin® and Levoleucovorin (Isovorin®), respectively (60 and 200 mg/m2).

ELIGIBILITY:
Main Inclusion Criteria:

* Operable colon cancer amenable to curative surgery.
* Performance status of 0 to 1
* Informed consent form
* Patients must be at least 18 years of age.

Main Exclusion Criteria:

* Any concurrent other anti-tumor therapy
* Any prohibited concomitant medication within 30 days of surgery
* Pregnancy or breast-feeding.
* Second primary malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Derwinger, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Levoleucovorin 200 mg/m2; Levoleucovorin 60 mg/m2: Levoleucovorin: i.v. bolus injection
- 6R-MTHF 200 mg/m2; 6R-MTHF 60 mg/m2: [6R] 5,10-methylenetetrahydrofolate: i.v. bolus injection
Period: Overall Study
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | 6R-MTHF 200 mg/m2 | 6R-MTHF 60 mg/m2
Started | 8 | 8 | 8 | 8
Completed | 8 | 7 | 8 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Modufolin 200 mg/m2; Modufolin 60 mg/m2: [6R] 5,10-methylenetetrahydrofolate: i.v. bolus injection
- Total: Total of all reporting groups
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 2 | 2 | 7
  >=65 years | 8 | 5 | 6 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.5 (9.15) | 66.71 (16.89) | 72 (15) | 71.75 (11.25) | 72.74 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 4 | 16
  Male | 4 | 3 | 5 | 4 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Concentration of [6R]-5,10-methylene-THF in Tumor Tissue
Description: Comparison of concentration of the active substance in Modufolin: [6R]-5,10-methylene-THF in tumor tissue after the different treatments.
Time Frame: Sample taken Day 1 (Day of surgery) at 0 min (before anesthetics) and 5, 10, 20, 40, 60, 90, 120, 180, 240, 360 min after study drug administration, and 24 h after study drug administration
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: pmol/g
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
pmol/g | 1871 (1159) | 959 (417) | 4725 (2210) | 2393 (1920)
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2 vs Modufolin 60 mg/m2; The exploratory evaluation of [6R]-5,10-methylene-THF concentration in tumor tissue was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0323, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1336, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8622, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0074, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2 vs Levoleucovorin 60 mg/m2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1752, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Concentration of [6R]-5,10-methylene-THF in Adjacent Mucosa Tissue
Description: Comparison of concentration of the active substance in Modufolin: [6R]-5,10-methylene-THF in mucosa adjacent to the tumor after the different treatments.
Time Frame: as for outcome 1
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: pmol/g
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
pmol/g | 1333 (852) | 626 (439) | 5099 (3927) | 3481 (3926)
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2 vs Modufolin 60 mg/m2; The exploratory evaluation of [6R]-5,10-methylene-THF concentration in mucosa adjacent to the tumor was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.1480, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0034, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0177, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0019, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2 vs Levoleucovorin 60 mg/m2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0118, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Concentration of [6S]-5-THF in Tumor Tissue
Description: Comparison of concentration of the metabolite [6S]-5-THF in tumor after the different treatments.
Time Frame: as for outcome 1
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: pmol/g
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
pmol/g | 1329 (720) | 933 (598) | 4175 (3127) | 2219 (1995)
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2 vs Modufolin 60 mg/m2; The exploratory evaluation of [6S]-5-THF concentration in tumor was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.1182, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0538, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5244, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0081, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0313, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2 vs Levoleucovorin 60 mg/m2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4777, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Concentration of [6S]-5-THF in Adjacent Mucosa Tissue
Description: Comparison of concentration of the metabolite [6S]-5-THF in mucosa adjacent to the tumor after the different treatments.
Time Frame: as for outcome 1
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: pmol/g
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
pmol/g | 1333 (852) | 626 (439) | 5099 (3927) | 3481 (3926)
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2 vs Modufolin 60 mg/m2; The exploratory evaluation of [6S]-5-THF concentration in mucosa adjacent to the tumor was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.2716, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0124, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0728, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0039, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2 vs Levoleucovorin 60 mg/m2; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0454, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Concentration of [6S]-5-methyl-THF in Tumor Tissue
Description: Comparison of concentration of the metabolite [6S]-5-methyl-THF in tumor after the different treatments.
Time Frame: as for outcome 1
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: pmol/g
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
pmol/g | 3574 (2415) | 1904 (918) | 4396 (1858) | 1882 (1204)
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2 vs Modufolin 60 mg/m2; The exploratory evaluation of [6S]-5-methyl-THF concentration in tumor was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0092, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.8303, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1182, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0081, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.3184, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2 vs Levoleucovorin 60 mg/m2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1752, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Concentration of [6S]-5-methyl-THF in Adjacent Mucosa Tissue
Description: Comparison of concentration of the metabolite [6S]-5-methyl-THF in mucosa adjacent to the tumor after the different treatments.
Time Frame: as for outcome 1
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: pmol/g
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
pmol/g | 3667 (2043) | 1216 (455) | 2494 (765) | 2066 (1517)
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2 vs Modufolin 60 mg/m2; The exploratory evaluation of [6S]-5-methyl-THF concentration in mucosa adjacent to the tumor was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0728, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.2246, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0428, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0003, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.4309, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2 vs Levoleucovorin 60 mg/m2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0055, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Concentration of [6S]-5-formyl-THF in Tumor Tissue
Description: Comparison of concentration of the metabolite [6S]-5-formyl-THF in tumor after the different treatments.
Time Frame: as for outcome 1
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: pmol/g
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
pmol/g | 3611 (3899) | 512 (259) | 100 (47) | 57 (48)
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2 vs Modufolin 60 mg/m2; The exploratory evaluation of [6S]-5-formyl-THF concentration in tumor was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0728, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0034, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0009, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2 vs Levoleucovorin 60 mg/m2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0055, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Concentration of [6S]-5-formyl-THF in Adjacent Mucosa Tissue
Description: Comparison of concentration of the metabolite [6S]-5-formyl-THF in mucosa adjacent to the tumor after the different treatments.
Time Frame: as for outcome 1
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: pmol/g
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
pmol/g | 5456 (3963) | 1403 (640) | 82 (77) | 42 (18)
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2 vs Modufolin 60 mg/m2; The exploratory evaluation of [6S]-5-formyl-THF concentration in mucosa adjacent to the tumor was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0240, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0058, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 60 mg/m2; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Levoleucovorin 200 mg/m2 vs Modufolin 200 mg/m2; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0014, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2 vs Levoleucovorin 60 mg/m2; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0338, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: AUC(0-2h) of [6R]-5,10-methylene-THF
Description: Area under the plasma concentration versus time curve from time 0 to 2 hours, for the active substance in Modufolin: [6R]-5,10-methylene-THF
Time Frame: Samples taken Day 1 (Day of surgery)
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: mcg*h/L
Groups:
- L-LV(200): Levoleucovorin 200 mg/m2
- L-LV(60): Levoleucovorin 60 mg/m2
- Mod(200): Modufolin 200 mg/m2
- Mod(60): Modufolin 60 mg/m2
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
mcg*h/L | 326.40261 (61.98416) | 239.90076 (0) | 7734.09113 (1557.76552) | 0 (0)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); The exploratory evaluation of AUC(0-2h) was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: AUC(0-2h) of [6S]-5-THF
Description: Area under the plasma concentration versus time curve from time 0 to 2 hours, for the metabolite [6S]-5-THF
Time Frame: Samples taken Day 1 (Day of surgery)
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: mcg*h/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
mcg*h/L | 827.1083 (178.23243) | 640.0489 (0) | 19408.1712 (3000.64794) | 5639.2700 (885.82223)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0009, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: AUC(0-2h) of [6S]-5-methyl-THF
Description: Area under the plasma concentration versus time curve from time 0 to 2 hours, for the metabolite: [6S]-5-methyl-THF
Time Frame: Samples taken Day 1 (Day of surgery)
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: mcg*h/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
mcg*h/L | 2336.24432 (829.18634) | 1258.60184 (247.51353) | 2277.89290 (1132.95603) | 997.74091 (413.68052)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0728, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.2246, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0166, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.1752, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.9581, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0118, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: AUC(0-2h) of [6SR]-5-formyl-THF
Description: Area under the plasma concentration versus time curve from time 0 to 2 hours, for the metabolite [6S]-5-formyl-THF
Time Frame: Samples taken Day 1 (Day of surgery)
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: mcg*h/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
mcg*h/L | 29911.9184 (6924.78031) | 7595.4599 (764.27650) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: AUC(Last) of [6R]-5,10-methylene-THF
Description: Area under the plasma concentration versus time curve, from time 0 to the last time point, for the active substance in Modufolin: [6R]-5,10-methylene-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: mcg*h/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
mcg*h/L | 462.10746 (221.85761) | 239.90076 (0) | 7910.61038 (1623.24300) | 2272.78010 (448.01407)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); The exploratory evaluation of AUC(last) was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0022, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: AUC(Last) of [6S]-5-THF
Description: Area under the plasma concentration versus time curve, from time 0 to the last time point, for the metabolite [6S]-5-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: mcg*h/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
mcg*h/L | 2231.1443 (1051.06650) | 640.0489 (0) | 28466.5389 (5303.28705) | 6766.9104 (1484.91243)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0009, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: AUC(Last) of [6S]-5-methyl-THF
Description: Area under the plasma concentration versus time curve, from time 0 to the last time point, for the metabolite [6S]-5-methyl-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: mcg*h/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
mcg*h/L | 32206.2771 (9121.1818) | 7689.0921 (5164.6098) | 21737.2428 (21757.1545) | 5495.1924 (6110.0065)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0240, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.1336, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.2725, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.1893, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: AUC(Last) of [6S]-5-formyl-THF
Description: Area under the plasma concentration versus time curve, from time 0 to the last time point, for the metabolite [6S]-5-formyl-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: mcg*h/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
mcg*h/L | 43429.1885 (12411.2844) | 9637.0308 (1637.2118) | 75.6174 (69.2176) | 50.1858 (0)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0142, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0085, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Cmax of [6R]-5,10-methylene-THF
Description: Maximum concentration (Cmax) in plasma of the active substance in Modufolin: [6R]-5,10-methylene-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
µg/L | 195.0000 (40.76763) | 123.0000 (0) | 22087.5000 (5635.45853) | 6452.8571 (559.18477)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); The exploratory evaluation of Cmax was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0014, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0021, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0014, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Cmax of [6S]-5-THF in Plasma
Description: Maximum concentration (Cmax) in plasma of the metabolite [6S]-5-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
µg/L | 577.6250 (190.74436) | 335.0000 (0) | 13372.5000 (2108.15932) | 5015.7143 (427.35064)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0009, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Cmax of [6S]-5-methyl-THF in Plasma
Description: Maximum concentration (Cmax) in plasma of the metabolite [6S]-5-methyl-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
µg/L | 2786.25000 (822.6253) | 1078.00000 (275.26206) | 2020.50000 (1142.25116) | 800.42857 (396.41849)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0240, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.1336, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.1551, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.1563, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Cmax of [6S]-5-formyl-THF in Plasma
Description: Maximum concentration (Cmax) in plasma of the active substance in Modufolin: [6R] 5,10- methylene-THF and the metabolites: [6S]-5-THF, [6S]-5-methyl-THF, and [6S]-5-formyl-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
µg/L | 32962.5000 (8594.17369) | 10168.3333 (2271.47896) | 252.7500 (141.51178) | 261.0000 (0)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0142, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0085, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Tmax of [6R]-5,10-methylene-THF
Description: Timepoint (tmax) when Cmax in plasma occurs of the active substance in Modufolin: [6R]-5,10-methylene-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 1.14285857 (0.53079605) | 1.00000000 (0) | 0.08333000 (0.00000000) | 0.08333000 (0.00000000)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); The exploratory evaluation of tmax was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0010, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0005, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Tmax of [6S]-5-THF
Description: Timepoint (tmax) when Cmax in plasma occurs for the metabolite [6S]-5-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 2.02083375 (1.03677360) | 1.50000000 (0) | 0.38541750 (0.24775936) | 0.09523571 (0.03149956)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0056, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0010, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0014, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Tmax of [6S]-5-methyl-THF
Description: Timepoint (tmax) when Cmax in plasma occurs for the metabolite [6S]-5-methyl-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 4.75000000 (1.38873015) | 2.41666667 (0.66458007) | 3.75000000 (1.16496475) | 2.92857143 (0.93222724)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.1796, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.3243, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0263, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0268, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.2041, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); Test type: Superiority; p = 0.0061, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Tmax of [6S]-5-formyl-THF
Description: Timepoint (tmax) when Cmax in plasma occurs for the metabolite [6S]-5-formyl-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 0.12499750 (0.08908753) | 0.08333000 (0.00000000) | 0.10416500 (0.04167000) | 0.08333000 (0)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: T(1/2) of [6R]-5,10-methylene-THF
Description: Terminal plasma elimination half-life time for the active substance in Modufolin: [6R]-5,10-methylene-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 3.07069184 (2.48958159) | 9.12204918 (0) | 0.90893994 (0.62586420) | 0.34368840 (0.06725217)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); The exploratory evaluation of t1/2 was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0268, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.0227, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.0933, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: T(1/2) of [6S]-5-THF
Description: Terminal plasma elimination half-life time for the metabolite [6S]-5-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 5.59459251 (1.76982092) | 0 (0) | 1.24808943 (0.23995973) | 0.96378070 (0.19174152)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.0177, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.0058, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.0043, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: T(1/2) of [6S]-5-methyl-THF
Description: Terminal plasma elimination half-life time for the metabolite [6S]-5-methyl-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 7.0955575 (1.18981597) | 10.7281060 (8.80812064) | 9.0743346 (3.84317226) | 8.5121573 (2.80644764)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: T(1/2) of [6S]-5-formyl-THF
Description: Terminal plasma elimination half-life time for the metabolite [6S]-5-formyl-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 1.51328500 (0.34108131) | 0.98944069 (0.20217367) | 0.23180085 (0.13438901) | 0 (0)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.0668, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.0502, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.0081, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: T(Last) of [6R]-5,10-methylene-THF
Description: The time-point for the last measurable concentration of the active substance in Modufolin: [6R]-5,10-methylene-THF
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 3.00000000 (1.41421356) | 2.00000000 (0) | 3.25000000 (1.38873015) | 1.35714286 (0.24397502)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); The exploratory evaluation of t(last) was done respectively for differences between treatments using Wilcoxon test. Differences in variability between the treatment groups were assessed using Proc GLM and Levene's test; Test type: Superiority; p = 0.0011, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.6691, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: T(Last) of [6S]-5-THF
Description: The time-point for the last measurable concentration for the metabolite [6S]-5-TH in plasma
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 4.75000000 (1.48804762) | 2.00000000 (0) | 5.75000000 (0.70710678) | 3.42857143 (0.78679579)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0015, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0640, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.1213, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: T(Last) of [6S]-5-methyl-THF
Description: The time-point for the last measurable concentration for the metabolite [6S]-5-methyl-THF in plasma
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 24.0000000 (0.00000000) | 12.0000000 (9.29516003) | 15.0000000 (9.62140471) | 8.5714286 (6.80336051)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.1791, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.4945, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0014, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.5990, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0303, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0107, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: T(Last) of [6S]-5-formyl-THF
Description: The time-point for the last measurable concentration for the metabolite [6S]-5-formyl-THF in plasma
Time Frame: Samples taken Day 1 (Day of surgery) and Day 2
Population: Per protocol population, all patients who complete the trial without any major deviations from the protocol procedure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | L-LV(200) | L-LV(60) | Mod(200) | Mod(60)
Number analyzed (Participants) | 8 | 6 | 8 | 7
h | 6.00000000 (0.00000000) | 8.33333333 (7.73735528) | 0.33333500 (0.23570226) | 0.16667000 (0)
Statistical Analysis 1: Comparison: Mod(200) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: L-LV(60) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: L-LV(200) vs Mod(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: L-LV(60) vs Mod(200); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0125, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: L-LV(200) vs Mod(200); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0017, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: L-LV(200) vs L-LV(60); [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.5286, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: Correlation Between Plasma and Tissue Concentration (Tumor and Mucosa) for [6R]-5,10-methylene-THF
Description: Correlation between the exposure of [6R]-5,10-methylene-THF following 2 hours after dosing (AUC[0-2h]) and the concentration of [6R]-5,10-methylene-THF in the tumor or adjacent mucosa at surgery.
Time Frame: Samples taken Day 1 (Day of surgery)
Population: The Per Protocol analysis set contained 29 of the 32 enrolled patients. One patient was withdrawn prior to study drug administration and two patients were excluded due to major protocol deviations.
Measure: Number; unit: correlation coefficient
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
correlation coefficient
  AUC(0-2h) vs. conc in tumor: number analyzed (Participants) | 7 | 1 | 8 | 0
  AUC(0-2h) vs. conc in tumor | 0.54039 | NA — Only one observation available for AUC(0-2h) | -0.21666 |
  AUC(0-2h) vs. conc in adjacent mucosa: number analyzed (Participants) | 7 | 1 | 8 | 0
  AUC(0-2h) vs. conc in adjacent mucosa | 0.68223 | NA — Only one observation available for AUC(0-2h) | 0.27618 |
Statistical Analysis 1: Comparison: Modufolin 200 mg/m2; AUC(0-2h) vs. concentration in tumor; Test type: Other; p = 0.6063, Pearson Correlation; Correlation factor = -0.21666
Statistical Analysis 2: Comparison: Levoleucovorin 200 mg/m2; AUC(0-2h) vs. concentration in tumor; Test type: Other; p = 0.2105, Pearson Correlation; Correlation factor = 0.54039
Statistical Analysis 3: Comparison: Modufolin 200 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.5079, Pearson Correlation; Correlation factor = 0.27618
Statistical Analysis 4: Comparison: Levoleucovorin 200 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.0913, Pearson Correlation; Correlation factor = 0.68223

34. Secondary Outcome: Correlation Between Plasma and Tissue Concentration (Tumor and Mucosa) for [6S]-5-THF
Description: Correlation between the exposure of [6S]-5-THF following 2 hours after dosing (AUC[0-2h]) and the concentration of [6S]-5-THF in the tumor or adjacent mucosa at surgery.
Time Frame: Samples taken Day 1 (Day of surgery)
Population: as for outcome 33
Measure: Number; unit: correlation coefficient
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
correlation coefficient
  AUC(0-2h) vs. conc in tumor | -0.02188 | NA — Only one observation available for AUC(0-2h) | 0.27018 | 0.38298
  AUC(0-2h) vs. conc in adjacent mucosa | 0.07937 | NA — Only one observation available for AUC(0-2h) | 0.34905 | 0.45404
Statistical Analysis 1: Comparison: Modufolin 60 mg/m2; AUC(0-2h) vs. concentration in tumor; Test type: Other; p = 0.3964, Pearson Correlation; Correlation factor = 0.38298
Statistical Analysis 2: Comparison: Modufolin 200 mg/m2; AUC(0-2h) vs. concentration in tumor; Test type: Other; p = 0.5175, Pearson Correlation; Correlation factor = 0.27018
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2; AUC(0-2h) vs. concentration in tumor; Test type: Other; p = 0.9590, Pearson Correlation; Correlation factor = -0.02188
Statistical Analysis 4: Comparison: Modufolin 60 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.3061, Pearson Correlation; Correlation factor = 0.45404
Statistical Analysis 5: Comparison: Modufolin 200 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.3967, Pearson Correlation; Correlation factor = 0.34905
Statistical Analysis 6: Comparison: Levoleucovorin 200 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.8518, Pearson Correlation; Correlation factor = 0.07937

35. Secondary Outcome: Correlation Between Plasma and Tissue Concentration (Tumor and Mucosa) for [6S]-5-methyl-THF
Description: Correlation between the exposure of [6S]-5-methyl-THF following 2 hours after dosing (AUC[0-2h]) and the concentration of [6S]-5-methyl-THF in the tumor or adjacent mucosa at surgery.
Time Frame: Samples taken Day 1 (Day of surgery)
Population: as for outcome 33
Measure: Number; unit: correlation coefficient
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
correlation coefficient
  AUC(0-2h) vs. conc in tumor | 0.73743 | 0.44757 | 0.03292 | 0.09033
  AUC(0-2h) vs. conc in adjacent mucosa | 0.76502 | 0.34496 | -0.66295 | 0.36854
Statistical Analysis 1: Comparison: Modufolin 60 mg/m2; AUC(0-2h) vs. conc in tumor; Test type: Other; p = 0.0586, Pearson Correlation; Correlation factor = 0.73743
Statistical Analysis 2: Comparison: Modufolin 200 mg/m2; AUC(0-2h) vs. conc in tumor; Test type: Other; p = 0.2661, Pearson Correlation; Correlation factor = 0.44757
Statistical Analysis 3: Comparison: Levoleucovorin 60 mg/m2; AUC(0-2h) vs. conc in tumor; Test type: Other; p = 0.9506, Pearson Correlation; Correlation factor = 0.03292
Statistical Analysis 4: Comparison: Levoleucovorin 200 mg/m2; AUC(0-2h) vs. conc in tumor; Test type: Other; p = 0.8315, Pearson Correlation; Correlation factor = 0.09033
Statistical Analysis 5: Comparison: Modufolin 60 mg/m2; AUC(0-2h) vs. conc in adjacent mucosa; Test type: Other; p = 0.0451, Pearson Correlation; Correlation factor = 0.76502
Statistical Analysis 6: Comparison: Modufolin 200 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.4027, Pearson Correlation; Correlation factor = 0.34496
Statistical Analysis 7: Comparison: Levoleucovorin 60 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.1513, Pearson Correlation; Correlation factor = -0.66295
Statistical Analysis 8: Comparison: Levoleucovorin 200 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.3690, Pearson Correlation; Correlation factor = 0.36854

36. Secondary Outcome: Correlation Between Plasma and Tissue Concentration (Tumor and Mucosa) for [6S]-5-formyl-THF
Description: Correlation between the exposure of [6S]-5-formyl-THF following 2 hours after dosing (AUC[0-2h]) and the concentration of [6S]-5-formyl-THF in the tumor or adjacent mucosa at surgery.
Time Frame: Samples taken Day 1 (Day of surgery)
Population: as for outcome 33
Measure: Number; unit: correlation coefficient
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
correlation coefficient
  AUC(0-2h) vs. conc in tumor: number analyzed (Participants) | 8 | 6 | 0 | 0
  AUC(0-2h) vs. conc in tumor | 0.68778 | 0.11512 |  |
  AUC(0-2h) vs. conc in adjacent mucosa: number analyzed (Participants) | 8 | 5 | 0 | 0
  AUC(0-2h) vs. conc in adjacent mucosa | 0.23512 | 0.02576 |  |
Statistical Analysis 1: Comparison: Levoleucovorin 200 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.5751, Pearson Correlation; Correlation factor = 0.23512
Statistical Analysis 2: Comparison: Levoleucovorin 60 mg/m2; AUC(0-2h) vs. concentration in adjacent mucosa; Test type: Other; p = 0.9672, Pearson Correlation; Correlation factor = 0.02576
Statistical Analysis 3: Comparison: Levoleucovorin 200 mg/m2; AUC(0-2h) vs. conc in tumor; Test type: Other; p = 0.0594, Pearson Correlation; Correlation factor = 0.68778
Statistical Analysis 4: Comparison: Levoleucovorin 60 mg/m2; AUC(0-2h) vs. conc in tumor; Test type: Other; p = 0.8281, Pearson Correlation; Correlation factor = 0.11512

37. Secondary Outcome: Gene Expression Ratios (Mucosa:Tumor)
Description: Concentration of different genes involved in folate transport and metabolism were analysed in both tumor and adjacent mucosa. The concentration in mucosa was divided by the concentration in tumor. A value above 1 indicate that the gene expression was higher in mucosa than in tumor and a value below 1 that the gene expression was higher in tumor than in mucosa.
Time Frame: Sample taken Day 1 (Day of Surgery)
Population: as for outcome 33
Measure: Number; unit: Ratio
Arm/Group | Modufolin 60 mg/m2 | Modufolin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Levoleucovorin 200 mg/m2
Number analyzed (Participants) | 7 | 8 | 6 | 8
Ratio
  AMT | 1.35 | 5.60 | 1.86 | 3.33
  PCFT | 2.03 | 2.75 | 2.92 | 2.45
  FPGS | 0.47 | 0.70 | 0.63 | 0.83
  MTHFS | 0.51 | 0.87 | 0.83 | 0.72
  ABCC3 | 1.83 | 3.37 | 2.48 | 4.15
  GGH | 0.50 | 0.47 | 0.35 | 0.31
  ABCC1 | 0.41 | 0.55 | 0.77 | 0.43
  MTHFD1L | 0.15 | 0.24 | 0.29 | 0.35
  SHMT1 | 0.89 | 1.13 | 0.72 | 2.26
  SHMT2 | 0.31 | 0.34 | 0.38 | 0.48
  RFC-1 | 0.48 | 0.66 | 0.53 | 1.18
Statistical Analysis 1: Comparison: Modufolin 60 mg/m2; Test type: Other; p = 0.0451, pearson

38. Secondary Outcome: Correlation of Gene Expression in Tumor and Adjacent Mucosa
Description: Concentration of the gene expression was analysed in both tumor and adjacent mucosa. The presence of any correlation between the results (i.e., concentration of the gene expression in tumor versus adjacent mucosa) was evaluated for each treatment. No evaluation was done between treatments.
Time Frame: Sample taken Day 1 (Day of Surgery)
Population: as for outcome 33
Measure: Number; unit: Normalized concentration
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
Normalized concentration
  AMT | -0.47193 | -0.70730 | 0.75404 | 0.42972
  PCFT | 0.11497 | 0.89976 | 0.58502 | 0.88128
  FPGS | 0.17664 | -0.64743 | 0.88682 | 0.97624
  MTHFS | 0.95840 | 0.58419 | 0.43194 | 0.94364
  ABCC3 | 0.00322 | 0.77700 | -0.25891 | -0.38987
  GGH | 0.78928 | -0.09737 | 0.46883 | 0.93711
  ABCC1 | 0.74757 | 0.14436 | -0.16724 | 0.82963
  MTHFD1L | 0.74459 | 0.20955 | 0.37160 | 0.32113
  SHMT1 | 0.59183 | 0.05531 | 0.67853 | 0.50966
  SHMT2 | 0.55508 | -0.71666 | 0.86266 | 0.81040
  RFC-1 | 0.64565 | -0.02450 | 0.23312 | 0.31800
Statistical Analysis 1: Comparison: Modufolin 60 mg/m2; Correlation for AMT gene expression; Test type: Other; p = 0.3359, Pearson Correlation; Correlation factor = 0.42972
Statistical Analysis 2: Comparison: Modufolin 200 mg/m2; Correlation for AMT gene expression; Test type: Other; p = 0.0307, Pearson Correlation; Correlation factor = 0.75404
Statistical Analysis 3: Comparison: Levoleucovorin 60 mg/m2; Correlation for AMT gene expression; Test type: Other; p = 0.1160, Pearson Correlation; Correlation factor = -0.70730
Statistical Analysis 4: Comparison: Levoleucovorin 200 mg/m2; Correlation for AMT gene expression; Test type: Other; p = 0.2377, Pearson Correlation; Correlation factor = -0.47193
Statistical Analysis 5: Comparison: Modufolin 60 mg/m2; Correlation for PCFT gene expression; Test type: Other; p = 0.0087, Pearson Correlation; Correlation factor = 0.88128
Statistical Analysis 6: Comparison: Modufolin 200 mg/m2; Correlation for PCFT gene expression; Test type: Other; p = 0.1277, Pearson Correlation; Correlation factor = 0.58502
Statistical Analysis 7: Comparison: Levoleucovorin 60 mg/m2; Correlation for PCFT gene expression; Test type: Other; p = 0.0146, Pearson Correlation; Correlation factor = 0.89976
Statistical Analysis 8: Comparison: Levoleucovorin 200 mg/m2; Correlation for PCFT gene expression; Test type: Other; p = 0.7863, Pearson Correlation; Correlation factor = 0.11497
Statistical Analysis 9: Comparison: Modufolin 60 mg/m2; Correlation for FPGS gene expression; Test type: Other; p = 0.0002, Pearson Correlation; Correlation factor = 0.97624
Statistical Analysis 10: Comparison: Modufolin 200 mg/m2; Correlation for FPGS gene expression; Test type: Other; p = 0.0033, Pearson Correlation; Correlation factor = 0.88682
Statistical Analysis 11: Comparison: Levoleucovorin 60 mg/m2; Correlation for FPGS gene expression; Test type: Other; p = 0.1645, Pearson Correlation; Correlation factor = -0.64743
Statistical Analysis 12: Comparison: Levoleucovorin 200 mg/m2; Correlation for FPGS gene expression; Test type: Other; p = 0.6756, Pearson Correlation; Correlation factor = 0.17664
Statistical Analysis 13: Comparison: Modufolin 60 mg/m2; Correlation for MTHFS gene expression; Test type: Other; p = 0.0014, Pearson Correlation; Correlation factor = 0.94364
Statistical Analysis 14: Comparison: Modufolin 200 mg/m2; Correlation for MTHFS gene expression; Test type: Other; p = 0.2852, Pearson Correlation; Correlation factor = 0.43194
Statistical Analysis 15: Comparison: Levoleucovorin 60 mg/m2; Correlation for MTHFS gene expression; Test type: Other; p = 0.2234, Pearson Correlation; Correlation factor = 0.58419
Statistical Analysis 16: Comparison: Levoleucovorin 200 mg/m2; Correlation for MTHFS gene expression; Test type: Other; p = 0.0002, Pearson Correlation; Correlation factor = 0.95840
Statistical Analysis 17: Comparison: Modufolin 60 mg/m2; Correlation for ABCC3 gene expression; Test type: Other; p = 0.3873, Pearson Correlation; Correlation factor = -0.38987
Statistical Analysis 18: Comparison: Modufolin 200 mg/m2; Correlation for ABCC3 gene expression; Test type: Other; p = 0.5358, Pearson Correlation; Correlation factor = -0.25891
Statistical Analysis 19: Comparison: Levoleucovorin 60 mg/m2; Correlation for ABCC3 gene expression; Test type: Other; p = 0.0691, Pearson Correlation; Correlation factor = 0.77700
Statistical Analysis 20: Comparison: Levoleucovorin 200 mg/m2; Correlation for ABCC3 gene expression; Test type: Other; p = 0.9940, Pearson Correlation; Correlation factor = 0.00322
Statistical Analysis 21: Comparison: Modufolin 60 mg/m2; Correlation for GGH gene expression; Test type: Other; p = 0.0018, Pearson Correlation; Correlation factor = 0.93711
Statistical Analysis 22: Comparison: Modufolin 200 mg/m2; Correlation for GGH gene expression; Test type: Other; p = 0.2413, Pearson Correlation; Correlation factor = 0.46883
Statistical Analysis 23: Comparison: Levoleucovorin 60 mg/m2; Correlation for GGH gene expression; Test type: Other; p = 0.8544, Pearson Correlation; Correlation factor = -0.09737
Statistical Analysis 24: Comparison: Levoleucovorin 200 mg/m2; Correlation for GGH gene expression; Test type: Other; p = 0.0199, Pearson Correlation; Correlation factor = 0.78928
Statistical Analysis 25: Comparison: Modufolin 60 mg/m2; Correlation for ABCC1 gene expression; Test type: Other; p = 0.0209, Pearson Correlation; Correlation factor = 0.82963
Statistical Analysis 26: Comparison: Modufolin 200 mg/m2; Correlation for ABCC1 gene expression; Test type: Other; p = 0.6922, Pearson Correlation; Correlation factor = -0.16724
Statistical Analysis 27: Comparison: Levoleucovorin 60 mg/m2; Correlation for ABCC1 gene expression; Test type: Other; p = 0.7850, Pearson Correlation; Correlation factor = 0.14436
Statistical Analysis 28: Comparison: Levoleucovorin 200 mg/m2; Correlation for ABCC1 gene expression; Test type: Other; p = 0.0330, Pearson Correlation; Correlation factor = 0.74757
Statistical Analysis 29: Comparison: Modufolin 60 mg/m2; Correlation for MTHFD1L gene expression; Test type: Other; p = 0.4825, Pearson Correlation; Correlation factor = 0.32113
Statistical Analysis 30: Comparison: Modufolin 200 mg/m2; Correlation for MTHFD1L gene expression; Test type: Other; p = 0.3647, Pearson Correlation; Correlation factor = 0.37160
Statistical Analysis 31: Comparison: Levoleucovorin 60 mg/m2; Correlation for MTHFD1L gene expression; Test type: Other; p = 0.6903, Pearson Correlation; Correlation factor = 0.20955
Statistical Analysis 32: Comparison: Levoleucovorin 200 mg/m2; Correlation for MTHFD1L gene expression; Test type: Other; p = 0.0341, Pearson Correlation; Correlation factor = 0.74459
Statistical Analysis 33: Comparison: Modufolin 60 mg/m2; Correlation for SHMT1 gene expression; Test type: Other; p = 0.2426, Pearson Correlation; Correlation factor = 0.50966
Statistical Analysis 34: Comparison: Modufolin 200 mg/m2; Correlation for SHMT1 gene expression; Test type: Other; p = 0.0643, Pearson Correlation; Correlation factor = 0.67853
Statistical Analysis 35: Comparison: Levoleucovorin 60 mg/m2; Correlation for SHMT1 gene expression; Test type: Other; p = 0.9171, Pearson Correlation; Correlation factor = 0.05531
Statistical Analysis 36: Comparison: Levoleucovorin 200 mg/m2; Correlation for SHMT1 gene expression; Test type: Other; p = 0.1222, Pearson Correlation; Correlation factor = 0.59183
Statistical Analysis 37: Comparison: Modufolin 60 mg/m2; Correlation for SHMT2 gene expression; Test type: Other; p = 0.0271, Pearson Correlation; Correlation factor = 0.81040
Statistical Analysis 38: Comparison: Modufolin 200 mg/m2; Correlation for SHMT2 gene expression; Test type: Other; p = 0.0058, Pearson Correlation; Correlation factor = 0.86266
Statistical Analysis 39: Comparison: Levoleucovorin 60 mg/m2; Correlation for SHMT2 gene expression; Test type: Other; p = 0.1090, Pearson Correlation; Correlation factor = -0.71666
Statistical Analysis 40: Comparison: Levoleucovorin 200 mg/m2; Correlation for SHMT2 gene expression; Test type: Other; p = 0.1533, Pearson Correlation; Correlation factor = 0.55508
Statistical Analysis 41: Comparison: Modufolin 60 mg/m2; Correlation for RFC-1 gene expression; Test type: Other; p = 0.4870, Pearson Correlation; Correlation factor = 0.31800
Statistical Analysis 42: Comparison: Modufolin 200 mg/m2; Correlation for RFC-1 gene expression; Test type: Other; p = 0.5785, Pearson Correlation; Correlation factor = 0.23312
Statistical Analysis 43: Comparison: Levoleucovorin 60 mg/m2; Correlation for RFC-1 gene expression; Test type: Other; p = 0.9632, Pearson Correlation; Correlation factor = -0.02450
Statistical Analysis 44: Comparison: Levoleucovorin 200 mg/m2; Correlation for RFC-1 gene expression; Test type: Other; p = 0.0838, Pearson Correlation; Correlation factor = 0.64565

39. Secondary Outcome: Homocystein Concentration
Description: Blood samples for folate biomarker (homocystein) analysis were collected at Screening, Day 2, and Day 5 (End of study visit).
Time Frame: Samples taken at Screening visit, Day 2, and End of Study (Day 5)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
μmol/L
  Concentration at Screening | 12.59 (4.28) | 11.27 (3.98) | 14.53 (6.22) | 13.80 (3.83)
  Concentration at Day 2 | 6.41 (2.32) | 6.40 (3.10) | 7.06 (1.97) | 8.14 (2.63)
  Concentration at Day 5 | 9.04 (2.53) | 9.18 (4.65) | 10.20 (3.34) | 10.10 (2.64)

40. Secondary Outcome: S-Folate Concentration
Description: Blood samples for folate biomarker (S-folate) analysis were collected at Screening, Day 2 and Day 5 (End of study visit).
Time Frame: Samples taken at Screening visit, Day 2 and End of Study (Day 5)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin 60 mg/m2
Number analyzed (Participants) | 8 | 6 | 8 | 7
nmol/L
  Concentration at Screening | 21.75 (8.88) | 21.00 (6.54) | 15.03 (5.20) | 18.71 (7.65)
  Concentration at Day 2 | 45.00 (0.00) | 45.00 (0.00) | 45.00 (0.00) | 45.00 (0.00)
  Concentration at Day 5 | 44.75 (0.71) | 40.80 (9.39) | 44.14 (2.27) | 40.29 (3.73)

41. Secondary Outcome: Change in Homocystein Concentration From Screening
Description: Blood samples for folate biomarker (homocystein) analysis were collected at Screening, Day 2 and Day 5 (End of study visit). Changes from screening to later visits were counted.
  The criteria for assessment categories "normal", "low" and "high" were based on the reference ranges for plasma-Homocystein as follows: "low" <4,7 mcmol/L; "normal" => 4,7 and <=16 mcmol/L; "high" >16 mcmol/L. Values were applicable for both male and female adults.
Time Frame: Samples taken at Screening visit, Day 2 and End of Study (Day 5)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Modufolin 60 mg/m2 | Modufolin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Levoleucovorin 200 mg/m2
Number analyzed (Participants) | 7 | 8 | 6 | 8
Participants
  Normal at Screen and Normal at Day 2 | 5 | 4 | 4 | 4
  Shift from Normal at Screen to Low at Day 2 | 0 | 1 | 2 | 2
  Shift from High at Screen to Normal at Day 2 | 2 | 3 | 0 | 2
  Normal at Screen and Normal at Day 5 | 5 | 5 | 4 | 6
  Shift from Normal at Screen to Low at Day 5 | 0 | 0 | 1 | 0
  Shift from High at Screen and Normal at Day 5 | 2 | 3 | 0 | 2
  Missing data Screen to Day 5 | 0 | 0 | 1 | 0

42. Secondary Outcome: Change in S-Folate Concentration From Screening
Description: Blood samples for folate biomarker (S-folate) analysis were collected at Screening, Day 2 and Day 5 (End of study visit). Changes from screening to later visits were counted.
Time Frame: Samples taken at Screening visit, Day 2 and End of Study (Day 5)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Modufolin 60 mg/m2 | Modufolin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Levoleucovorin 200 mg/m2
Number analyzed (Participants) | 7 | 8 | 6 | 8
Participants
  Shift from Normal at Screen to High at Day 2 | 7 | 8 | 5 | 8
  Missing data Screen to Day 2 | 0 | 0 | 1 | 0
  Normal at Screening and Normal at Day 5 | 3 | 1 | 1 | 0
  Shift from Normal at Screen to High at Day 5 | 4 | 6 | 4 | 8
  Missing data Screen to Day 5 | 0 | 1 | 1 | 0

43. Secondary Outcome: Number of AEs Per Severity
Description: Number of reported AEs per treatment with respect to severity
Time Frame: Screening visit until end of study, Day 5
Population: The safety population contained 31 of the 32 enrolled patients. One patient randomized to L-LV 60 mg/m2 was withdrawn prior to study drug administration and thus excluded from the safety analysis set.
Measure: Number; unit: Events
Groups:
- Modufolin mg/m2: [6R] 5,10-methylenetetrahydrofolate: i.v. bolus injection
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | Modufolin 200 mg/m2 | Modufolin mg/m2
Number analyzed (Participants) | 8 | 7 | 8 | 8
Events
  AEs of mild severity | 1 | 0 | 1 | 5
  AEs of moderate severity | 3 | 0 | 7 | 2
  AEs of severe severity | 0 | 1 | 2 | 2

ADVERSE EVENTS:
Arm/Group | Levoleucovorin 200 mg/m2 | Levoleucovorin 60 mg/m2 | 6R-MTHF 200 mg/m2 | 6R-MTHF 60 mg/m2
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/7 | 2/8 | 2/8
Other Adverse Events (participants affected / at risk) | 4/8 | 2/7 | 4/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levoleucovorin 200 mg/m2 (N=8) | Levoleucovorin 60 mg/m2 (N=7) | 6R-MTHF 200 mg/m2 (N=8) | 6R-MTHF 60 mg/m2 (N=8)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute mycardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levoleucovorin 200 mg/m2 (N=8) | Levoleucovorin 60 mg/m2 (N=7) | 6R-MTHF 200 mg/m2 (N=8) | 6R-MTHF 60 mg/m2 (N=8)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other